CLINICAL TRIAL: NCT03509844
Title: Comparison of Treatments for Complex Posttraumatic Stress Disorder -a Randomized Controlled Trial
Brief Title: The Modum Bad Complex Posttraumatic Stress Disorder Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modum Bad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPTSD-Peter_Sele
Record Dates: First submitted 2018-03-22; First posted 2018-04-26 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome is assessed with CAPS-V by research assistants blind to the patients allocation to treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prolonged Exposure (Experimental): Psychotherapy: 10 weeks, Prolonged Exposure (individual sessions) according to the manual developed by Foa et al., adapted for a residential care setting
  Interventions: Behavioral: Psychotherapy
- STAIR (Experimental): Psychotherapy: 10 weeks, Skills Training in Affect and Interpersonal Regulation (STAIR) (group sessions), according to the manual developed by Cloitre et al., adapted for a residential care setting
  Interventions: Behavioral: Psychotherapy
- STAIR/NT (Experimental): Psychotherapy: 16 weeks, 10 weeks Skills Training in Affect and Interpersonal Regulation (STAIR) (group sessions), followed by 6 weeks of Narrative Therapy (NT) (individual sessions), according to the manual developed by Cloitre et al., adapted for a residential care setting.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Three established psychotherapeutic models for treatment of complex posttraumatic stress disorders are compared in a residential care setting. Combination of group and individual sessions.

SUMMARY:
This study compares three established, manual based psychotherapies for Complex Post-traumatic Stress disorder (CPTSD) in patients with childhood trauma (e.g. sexual abuse, violence). The primary aim of the study is to compare phase-oriented treatment (Stabilization + Exposure) with two non-phased treatments, Exposure and Stabilization.

DETAILED DESCRIPTION:
Available treatment procedures for PTSD are largely developed within the context of adult trauma (e.g. accidents, natural disasters, rape or combat). The need for additional treatment options targeting dysfunctional affect regulation and interpersonal problems in patients suffering after childhood trauma is debated in research and clinical settings.

96 patients will be recruited from referrals to an in-patient clinic in Norway called Modum Bad. After assessment, patients will be randomly assigned to one of three treatment arms. One-third will receive 10 weeks of Prolonged Exposure, one-third 10 weeks of Skills Training in Affect and Interpersonal Regulation (STAIR), and the last third a phase-based treatment lasting 16 weeks (STAIR + Narrative Therapy).

ELIGIBILITY:
Inclusion Criteria:

* childhood trauma (e.g. sexual abuse, violence prior to age 18),
* a diagnosis of Posttraumatic Stress Disorder PTSD according to DSM-5
* a diagnosis of Complex PTSD according to the suggested additional criteria for complex PTSD in International Classification of Diseases (ICD-11)

Exclusion Criteria:

* severe psychotic disorder
* dissociative identity disorder (DID)
* active phase substance dependence
* acute suicidality
* major current life crisis
* severely disturbed group functioning
* mental disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS-5) for the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) | approximately 15 months
  30 items structured interview corresponding to the definition of PTSD in DSM-5. 20 items correspond to the symptoms for PTSD and are scored on a 0-4 severity scale to establish symptom severity (range 0-40)

SECONDARY OUTCOMES:
The PTSD Checklist for DSM-5 (PCL-5) | approximately 15 months
  20 items self-report measure for PTSD symptoms corresponding to DSM-5 criteria for PTSD. Severity is scored on a 0-4 scale (range 0-40)
Inventory of Interpersonal Problems (IIP-64) | approximately 15 months
  64 items self-report measure for interpersonal problems. Severity is scored on a 0-4 scale (range 0-256)
Beck Depression Inventory-Second Edition (BDI-II) | approximately 15 months
  21 item self-report measure for depressive symptoms. Severity is scored on a 0-3 scale (range 0-63

CONTACTS AND LOCATIONS:
Locations (1):
- Modum Bad, Vikersund, Buskerud, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sele P, Hoffart A, Cloitre M, Hembree E, Oktedalen T. Comparing phase-based treatment, prolonged exposure, and skills-training for Complex Posttraumatic Stress Disorder: A randomized controlled trial. J Anxiety Disord. 2023 Dec;100:102786. doi: 10.1016/j.janxdis.2023.102786. Epub 2023 Oct 12. PMID 37871452